CLINICAL TRIAL: NCT05272566
Title: Prephage - Faecal Bacteriophage Transfer for Enhanced Gastrointestinal Tract Maturation in Preterm Infants - Donor Study
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Lise Aunsholt, Neonatologist, Clinical Professor (Unknown)
Responsible Party: Principal Investigator, Gustav Riemer Jakobsen, Medical Doctor, Ph.d-student, Rigshospitalet, Denmark
Other Study IDs: PrePhage, Donor
Record Dates: First submitted 2022-02-15; First posted 2022-03-09 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Feeding Patterns; Microbial Colonization
Keywords: Microbiome; Bacteriophage; Feeding Pattern; Stool Pattern
MeSH Terms: conditions — Feeding Behavior; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal Samples from both mothers and infants, only non-human DNA/RNA analyzed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infants: 30 healthy, term infants are recruited for 2 purposes:
  1. To study the development of gut bacteria and viruses over time
  2. To use as donors in a separate trial
- Mothers: 30 healthy pregnant women are recruited along with their infants
  1. To compare gut bacteria and viruses with those of their children
  2. To screen for disease transferrable by breastfeeding

SUMMARY:
PrePhage - Fecal bacteriophage transfer for enhanced gastrointestinal tract maturation in preterm infants

This pilot triol has the primary goal of demonstrating the safety of transferring viruses and proteins from healthy term infants to preterm infants born between gestational age (GA) 26 + 0 and 30+6. The long-term goal is to develop a safe and effective treatment to prevent the severe gut disease called necrotizing enterocolitis (NEC).

NEC is a common disease in neonatal intensive care units affecting 5-10% of all admitted patients. 15-30% of the affected children die from the disease, and many of the survivors suffer from the effects of extensive gut surgery.

While the disease is caused by many different factors, recent research has shown the gut microbiome to be a central factor in the development of NEC. Furthermore, in the recent years special viruses called bacteriophages have shown potential in the treatment of various diseases.

By collecting feces from healthy, term infants and filtering it thoroughly, the investigators can provide a treatment that contains practically only viruses, proteins and nutrients. It is our belief that giving the preterm infants a mix of viruses including bacteriophages will prevent NEC.

To do this, the investigators will go through 3 stages:

Recruiting and following healthy donor infants to study the microbiota and use feces from them to donate in stage 2 and 3 Examining the safety of the treatment as well as how it works in preterm piglets

STAGE 3 will be performed only if stage 2 shows no serious risks for the infants

Testing the treatment in preterm infants. 10 preterm infants will receive the treatment and 10 preterm infants will receive placebo. The investigators expect to see no serious side effects to the treatment. The investigators hope, but do not expect to be able to see a beneficial effect of the treatment.

If this pilot trial shows promising results, it will be followed be a larger clinical trial.

DETAILED DESCRIPTION:
Detailed Description:

PrePhage - Fecal bacteriophage transfer for enhanced gastrointestinal tract maturation in preterm infants

This pilot trial aims to investigate if fecal filtrate transfers (FFT) to preterm infants is safe and tolerable. To investigate this, the investigators will recruit 20 donor infants and their mothers from time of delivery, and both will be subjected to a novel screening program including blood, urine, breastmilk, fecal screening and standard clinical investigation. Donor fecal samples will be collected from time of birth and with varying intervals for consecutive 3 years for 3 purposes: 1) to conduct safety studies in preterm piglets before transfer to preterm recipient infants, 2) to conduct FFT to preterm infants, and 3) to map normal microbiota development in healthy infants. The feces used for donation will be collected between 2-4 weeks after birth. After 1 year, donated feces will be released for FFT to preterm, but only if the donor infant at this time has been healthy and normally developed. Donors are followed up for consecutive 3 years after birth. Maternal fecal samples will be compared to infant samples, to investigate maternal to infant transfer of microbiota, as well as changes in infant microbiota in response to environment.

20 preterm infants with gestational age between 26 +0 - 30+6 weeks + days, are block randomized to either FFT or saline placebo within 24 hours after birth and the following 3 days, in total 4 donations. The recipients are clinically and biochemically closely monitored by attending staff and the group of investigators according to best clinical practice and predefined clinical observation. The recipients are followed up for consecutive 3 years to evaluate potential late side-effects and to monitor change in fecal microbiome after transplant or placebo.

The primary endpoint is to assess safety of FFT to preterm infants with expected no increase in necrotizing enterocolitis (NEC), sepsis and death in the intervention group. The secondary endpoint is to assess if, FFT treatment will reduce incidence of feeding tolerance and improve healthy gut development in recipient preterm infants. The investigators expect to find FFT safe and with fewer cases of NEC and sepsis. The investigators do not expect to prove the effect of the intervention in this study. However, the investigators aim to follow up with a double-blinded multicenter randomized control trial - powered to document our hypothesis - that when colonizing with a healthy microbiome, it is possible decrease incidence of NEC in premature infants.

ELIGIBILITY:
Inclusion criteria for infants

* The donor must be of term (>37+0 weeks GA, < 41+0 weeks GA),
* Be born vaginally with no maternal pre-birth infection,
* Be exclusively breastfed un till fulfilled donation at 4 weeks of age,
* Have no known predisposition for disease.

Exclusion criteria for infants

* Antibiotic exposure before collection of faecal material for donation,
* Disease between time of birth and collection of feces for donation,
* Major congenital anomalies or birth defects, perinatal asphyxia, need for mechanical ventilation or cardiovascular support before time of inclusion.
* Positive stool sample for C. difficile toxin, parasites or other pathogens
* Positive HIV, HBV, or HCV or CMV
* Parents who do not want to know the HIV, HBV or HCV status of the child

Inclusion criteria for mothers

* Women aged 18-45 and currently healthy
* No continuous medical consumption with effects on microbiome
* Non-smoking
* Ability to give informed consent

Exclusion criteria for mothers

* Known or high risk of infectious disease such as HIV, HBV, or HCV
* Positive CMV IgM during pregnancy
* Positive stool sample for C. difficile toxin, parasites or other pathogens
* Systemic antibiotic treatment < 1 months prior to study
* New tattoo < 1 month prior to study
* Risky sexual behavior
* Gestational diabetes
* Family history of inflammatory bowel disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Families are recruited from out-patients clinics at the secondary level in Copenhagen
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Gut microbiome | 1 year
  Total genomic DNA will be subjected to deep metagenome sequencing and related to the study outcomes. When extracting faecal DNA as well as viral DNA/RNA, physical fractionation or selective lysis will be employed to ensure host DNA is kept to a minimum. Remaining host DNA material will be removed during bioinformatics filtering and mapping of the shotgun metagenomics data.

SECONDARY OUTCOMES:
Clinical development | 1 year
  Clinical evaluation by pediatric doctor, outcome is dichotomous in terms of following normal development or not according to clinical evaluation
Weight | 1 year
  weight in kilograms
Length | 1 year
  Length in centimeters
Time to establish breastfeeding | 2 weeks
  Days from birth till sufficiently breastfeeding
Length of hospital stay after birth | 1 month
  Length of hospital stay after birth
Days to regain birthweight | 1 month
  Time after birth to regain birthweight
Stool characteristics - Amount | 1 year
  Score from 1-4 using Amsterdam Stool Scale
Stool characteristics - Consistency | 1 year
  Score from 1-6 using Diapered Infant Stool Scale
Stool characteristics - Color | 1 year
  Score from 1-6 using Amsterdam Stool Scale
Defacation frequency | 1 year
  Amount af defacations per week
Full solid food | 1 year
  Age at which infant is no longer breastfed
Frequency of infections | 1 year
  Infections per year

CONTACTS AND LOCATIONS:
Overall Officials: Lise Aunsholt, md, phd, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Gustav R Jakobsen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Truly anonymizing data with infants recently born in a small society such as Denmark is challenging. The data may be released at a later date.

REFERENCES:
- [Derived] Kappel SS, Jakobsen GR, Oestergaard KL, Brunse A, Nielsen DS, Aunsholt L. Parental Consent to a Neonatal Clinical Study: The Roles of Uncertainty, Burden of Sample Collection and Societal Expectations. Acta Paediatr. 2025 Oct 6. doi: 10.1111/apa.70333. Online ahead of print. PMID 41051016

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT05272566/Prot_SAP_000.pdf